CLINICAL TRIAL: NCT05670119
Title: The Effect of Catheter-Associated Infection Control Training on Surgical Nurses' Knowledge and Attitude Levels
Brief Title: The Effect of Catheter-Associated Infection Control Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-245
Record Dates: First submitted 2022-12-19; First posted 2023-01-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Infection Control Training
Keywords: Attitude, Infection, Knowledge, Surgical Nursing
MeSH Terms: conditions — Behavior; Infections

STUDY DESIGN:
Intervention Model Description: This study is a single-center parallel-group randomized controlled clinical trial. Participants who accepted to participate in the study and met the inclusion criteria will be assigned to the intervention (n=35) or control group (n=35) according to the computer-based randomization table.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Nurses in the intervention group will be given face-to-face training on evidence-based catheter-related infection control measures. The content of the training program will also be given to the participants as written material (brochure). The training will take an average of 30 minutes. After the data collection forms are applied to the participants in the intervention group (pre-test), evidence-based training on catheter-related infection control measures will be conducted. The forms will be applied again immediately after the training (post-test) to measure the knowledge level of nurses and three months after the training (post-test) to measure the level of attitude.
  Interventions: Other: Structured Training
- Control Group (No Intervention): Routine in-service training practices will be given to the control group. Data collection forms will be applied to the participants in the control group at the same time as the intervention group.

INTERVENTIONS:
Other: Structured Training — Structured catheter-related infection control training was prepared by using evidence-based information and receiving 10 expert opinions. This training will be given to the participants with a face-to-face PowerPoint presentation by the infection control nurse (researcher) and will also be presented as written material.
  Arms: Intervention Group

SUMMARY:
The goal of this type of study: clinical trial is to determine the effectiveness of educational practices on catheter-associated infection control measures on surgical nurses. The main question it aims to answer are:

* Is there a difference between the knowledge and attitude levels of surgical nurses receiving and not receiving catheter-related infection control training on preventing peripheral and central catheter-related bloodstream infections?
* Is there a difference between the knowledge and attitude levels of surgical nurses receiving and not receiving catheter-related infection control training to prevent catheter-related urinary tract infections?

The main tasks that the participants will be asked to do will be explained and their consent will be obtained. The two research groups will be compared.

DETAILED DESCRIPTION:
This study will be conducted with a total of 70 nurses working in the surgical clinics of a city hospital in Istanbul and meeting the inclusion criteria. Nurses who meet the inclusion criteria of the study will be divided into two groups: intervention (n=35) and control group (n=35) according to the randomization method created with computer-based random numbers. Nurses in the intervention group will be given face-to-face training on evidence-based catheter-related infection control measures. The content of the training program will also be given to the participants as written material (brochure). The training will take an average of 30 minutes. Routine in-service training practices will be given to the control group. Descriptive Characteristics Form, the Peripheral and Central Venous Catheter-Related Bloodstream Infection Prevention Knowledge and Attitudes Scale, and Catheter-Associated Urinary Tract Infections Control Precautions will be used in data collection. Data will be collected from all participants before, immediately after, and three months after the training practices.

ELIGIBILITY:
Inclusion Criteria:

* Being a nurse
* Working in the surgical unit
* Agreeing to participate in the research

Exclusion Criteria:

* Being on leave/reported (maternity leave, unpaid leave, medical report, etc.)
* Not filling out the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The peripheral and central venous catheter-related bloodstream infection prevention knowledge and attitudes of the surgical nurses" | 0-3 months
  There is a difference between 0-3 months on the knowledge and attitudes of the training given to nurses to prevent peripheral and central venous catheter-related bloodstream infections. The Peripheral and Central Venous Catheter-Related Bloodstream Infection Prevention Knowledge and Attitudes Scale will be administered to the all participants before the training (pre-test). This scale will be used again immediately after the training (post-test) to measure the knowledge level of nurses and three months after the training (post-test) to measure the level of attitude. The scale includes 14 items and consists of "general precautions" and "catheter care" sub-dimensions. The scale score range is 14-70 points. Higher scores on the scale indicates higher knowledge and attitude.
The catheter-associated urinary tract infections control precautions knowledge and attitudes of the surgical nurses | 0-3 months
  There is a difference between 0-3 months on the knowledge and attitudes of the training given to nurses to prevent catheter-associated urinary tract infections. The Catheter-Associated Urinary Tract Infections Control Precautions Scale will be administered to the all participants before the training (pre-test). This scale will be used again immediately after the training (post-test) to measure the knowledge level of nurses and three months after the training (post-test) to measure the level of attitude. The scale includes 15 items and consists of "standard precautions", "maintenance of the closed drainage system" and "catheter-bag change" sub-dimensions. The scale score range is 15-75 points. Higher scores on the scale indicates higher knowledge and attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Filiz Akdemir, RN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Habibe Filiz Akdemir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakan AB, Arli SK. Development of the peripheral and central venous catheter-related bloodstream infection prevention knowledge and attitudes scale. Nurs Crit Care. 2021 Jan;26(1):35-41. doi: 10.1111/nicc.12422. Epub 2019 Feb 28. PMID 30815969
- [Background] Suha BK, Karagozoglu S. The Effect of a Guide Based Application Bundle on the Catheter-Related Infection. Florence Nightingale Hemsire Derg. 2019 Oct 1;27(3):222-230. doi: 10.5152/FNJN.2019.426870. eCollection 2019 Oct. PMID 34267976
- See also: Guideline for Hand Hygiene in Health-Care Settings Recommendation of the Healthcare Infection Control Practices Advisory Committee and the HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. — http://www.cdc.gov/mmwr/pdf/rr/rr5116.pdf
- See also: Bloodstream infection event (Central line-associated bloodstream ınfection and non-central line associated bloodstream infection). — http://www.cdc.gov/nhsn/pdfs/pscmanual/4psc_clabscurrent.pdf
- See also: Healthcare associated infections acquired in intensive care units - annual epidemiological report for 2015. Stockholm (Sweden): European Centre for Disease Prevention and Control. — http://www.ecdc.europa.eu/sites/default/files/documents/AER_for_2015-healthcare-associated-infections_0.pdf